CLINICAL TRIAL: NCT03308032
Title: Self-Directed Online Training for Chinese Caregivers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Environment and Health Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NIH 1R43HL115924-01
Record Dates: First submitted 2017-10-03; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Dementia; Alzheimer Disease
MeSH Terms: conditions — Dementia; Alzheimer Disease | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants assigned to the intervention arm will be invited to connect to a webpage, through either computer or tablet / iPad, where they can login to receive the SDL course. Immediately after the login, and weekly thereafter, participants will receive emails to remind them of the login passwords, to provide them with tracking data on their progress in going through the training lessons. For those who login but do not proceed to take baseline assessment for longer than two days, study staff will contact participants, via the email address or telephone number that was entered during initial registration for login, to answer any questions they might have and to provide assistance to those who have not been able to log onto the site. Those who sign up without taking any courses for 10 days will receive a reminder call by study staff. Intervention arm participants will be invited back via both
  Interventions: Behavioral: Intervention
- Control (Active Comparator): Participants assigned to the intervention arm will be invited to connect to a webpage, through either computer or tablet / iPad, where they can login to receive the SDL course.
  Immediately after the login, and weekly thereafter, participants will receive emails to remind them of the login passwords, to provide them with tracking data on their progress in going through the training lessons (see below). For those who login but do not proceed to take baseline assessment for longer than two days, study staff will contact participants, via the email address or telephone number that was entered during initial registration for login, to answer any questions they might have and to provide assistance to those who have not been able to log onto the site. Those who sign up without taking any courses for 10 days will receive a reminder call by study staff. Intervention arm participants will be invited back via both
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention — SDL intervention employs a comprehensive engagement design that includes seven innovative strategies: 1) customization of content of the training curriculum to fit individual learner's needs; 2) tailoring the length of trainings by using short video clips to allow caregivers flexibility in completing the curriculum; 3) using an instructional format (SCHOLAR) designed to maximize active learning during each training lesson; 4) progress tracking to help the learner stay focused and motivated; 5) a recommendation algorithm that facilitates the learner's transition from one training topic to the next; 6) behavioral economics-based messages, to re-engage the learner if he/she stops participating
  Arms: Intervention
Behavioral: Control — Participants in the control group will be invited to a comparable online training course consisting of all of our training video clips, without the interactive engagement design features. These represent standard video training based on evidence-based content.
  Arms: Control

SUMMARY:
The proposed project seeks to develop an online self-directed learning (SDL) intervention program that seeks to improve caregiving and self-care skills among ethnic Chinese dementia caregivers. The benefits of such a product may include improved psychological health in caregivers and a reduction in behavioral disturbances among elderly care recipients with dementia.

DETAILED DESCRIPTION:
The objective of this Phase II application is to develop an online self-directed learning (SDL) intervention program that seeks to improve caregiving and self-care skills among ethnic Chinese dementia caregivers. The benefits of such a product may include improved psychological health in caregivers and a reduction in behavioral disturbances among elderly care recipients with dementia. While online dementia caregiver interventions are advantageous in reaching broad audiences, these individuals face significant challenges in engaging the target audience and keeping them engaged throughout the intervention program. The proposed online SDL skill training intervention addresses these challenges with a comprehensive engagement design to ensure retention and effective learning in the training program.

All Phase I Study Aims have been successfully completed. The prototype provides preliminary evidence that an SDL training intervention is able to successfully engage ethnic Chinese caregivers of elders with dementia, improving perceived self-efficacy to manage caregiving tasks, while reducing negative emotions in the caregiver. Phase II Specific Aims: The Phase II study will further develop the prototype into a fully-functioning online SDL skill training intervention for ethnic Chinese dementia caregivers, and evaluate it in a randomized control trial. In Specific Aim 1, the research team will develop additional multi-lingual training video clips to complete the training program, and make them available for Cantonese-, Mandarin-, and/or English-speaking caregivers from different Chinese cultural backgrounds. In Specific Aim 2, the research team will develop software that enables and integrates all engagement design functionalities. In Specific Aim 3, the research team will conduct a randomized controlled trial to evaluate the effectiveness of the SDL training intervention based on a comprehensive engagement design (intervention arm) compared to one that does not rely on a comprehensive engagement design (control arm).

Evidence of the effectiveness of the SDL intervention will contribute to the larger information and communication technology field, increasing the public's understanding and basic knowledge of effective engagement in the rapidly growing field of online health interventions. The comprehensive engagement approach developed through this research could be transferred to other ethnic minority groups facing dementia caregiving challenges, as well as other populations facing challenges related to the management of other chronic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Ethnic Chinese Caregiver

Exclusion Criteria:

* Not Chinese or Caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-03-05 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in Stress Level | At Week 1 and at Week 12
  Will be assessed using the 10 point Perceived Stress Scale